CLINICAL TRIAL: NCT03070912
Title: Study of the Frequency of Hemorrhages Associated With the Functional Anomalies of Willebrand Factor in Emergency Patients of a Veino Arterial or Veinous ECMO
Brief Title: Frequency of Hemorrhages Associated With the Functional Anomalies of Willebrand Factor in Emergency Patients
Acronym: WITECMO-H
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_83; 2017-A00256-47 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-02-13; First posted 2017-03-06 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Von Willebrand Diseases
Keywords: mechanical circulatory support; bleeding, acquired von willebrand disease; acquired von willebrand disease
MeSH Terms: conditions — von Willebrand Diseases; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ECMO has improved the outcome of heart or respiratory failure and carcinogenic shock and are increasingly used. However bleeding complications occurring in up to 50% of patients are poorly understood and worsen the overall results. The aim is to investigate the occurence of bleeding and its frequency according to the type of ECMO either veno-arterial or veno-venous. The investigators also want to assess the relation of bleeding with von Willebrand Factor defects.

ELIGIBILITY:
Inclusion Criteria:

* informed consent of patient or person in charge
* patient supplied by an ECMO for cardiac or respiratory failure and referred to Lille University Hospital
* patient affiliated to "french social security"

Exclusion Criteria:

* pregnant woman
* no consent
* no affiliation to
* patient affiliated to '
* preexisting bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients older than 18 years receiving either veno-arterial or even-venous ECMO and referred at Lille University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of major bleeding | During ECMO support, up to 3 weeks after implantation
  Number of major bleeding events (BARC classification ) occurring within the time course of support by ECMO

SECONDARY OUTCOMES:
Number of Participants With Abnormal VWF functional activities and multimeric profile according to the type of ECMO support (VA- or VV-ECMO) | 1 hour, 24 hours and day seven after implantation
  Willebrand Factor abnormalities according to the type of ECMO support (VA- or VV-ECMO)
Number of Participants With Abnormal VWF functional activities and multimeric profile before and after the first reduction in VA-ECMO flow rate | During ECMO support, up to 3 weeks after implantation
  Willebrand Factor abnormalities according to residual arterial pulsatility levels under VA-ECMO
Number of Participants With Abnormal VWF functional activities and multimeric profile in 2 groups defined by the level of pulse pressure measured before ECMO weaning: high (> median) or low (< median) pulse pressure | During ECMO support, up to 3 weeks after implantation
  Willebrand Factor abnormalities according to residual arterial pulsatility levels under VA-ECMO
Number of Participants With major bleeding events (BARC classification) before and after the first reduction in VA-ECMO flow rate | During ECMO support, up to 3 weeks after implantation
  Willebrand Factor abnormalities according major bleeding events under VA-ECMO
Number of Participants With major bleeding events (BARC classification) in 2 groups defined by the level of pulse pressure measured before ECMO weaning: high (> median) or low (< median) pulse pressure | During ECMO support, up to 3 weeks after implantation
  Willebrand Factor abnormalities according major bleeding events under VA-ECMO
Frequency of major bleeding events according to diabetes status | During ECMO support, up to 3 weeks after implantation
  Number of major bleeding events (BARC classification ) occurring within the time course of support by ECMO in patients with and without diabetes
Frequency of major thrombotic events according to diabetes status | During ECMO support, up to 3 weeks after implantation
  Number of major thrombotic events (stroke, transient ischemic attack, acute limb ischemia, ECMO thrombosis) occurring within the time course of support by ECMO in patients with and without diabetes
Frequency of pro-thrombotic biological abnormalities | During ECMO support, up to 3 weeks after implantation
  Measurement of plasma free hemoglobin, leuco-platelet aggregates and neutrophil extracellular traps levels

CONTACTS AND LOCATIONS:
Overall Officials: Antoine RAUCH, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - CH ARRAS, Arras
  - CH Boulogne, Boulogne-sur-Mer
  - CH DOUAI, Douai
  - CH Dunkerque, Dunkirk
  - Hôpital Cardiologie, CHU, Lille
  - Ch Tourcoing, Tourcoing
  - Ch Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moussa MD, Abou-Arab O, Staessens S, Jungling M, Labreuche J, Lamer A, Beyls C, Rousse N, Rauch A, Loobuyck V, Beaudeux C, Pierache A, Deblauwe D, Corseaux D, Dubernet M, Guilbart M, Thellier L, Mahjoub Y, Juthier F, Dupont H, De Meyer SF, Vincentelli A, Susen S, Robin E. Comparison of the effects of phosphorylcholin versus heparin-based surface coating on clinical and histologic outcomes during veno-arterial extracorporeal membrane oxygenation support: a propensity score weighted analysis. J Thromb Haemost. 2025 Jun;23(6):1879-1892. doi: 10.1016/j.jtha.2025.02.020. Epub 2025 Feb 26. PMID 40020783
- [Result] Rauch A, Dupont A, Rosa M, Desvages M, Le Tanno C, Abdoul J, Didelot M, Ung A, Ruez R, Jeanpierre E, Daniel M, Corseaux D, Spillemaeker H, Labreuche J, Pradines B, Rousse N, Lenting PJ, Moussa MD, Vincentelli A, Bordet JC, Staels B, Vincent F, Denis CV, Van Belle E, Casari C, Susen S. Shear Forces Induced Platelet Clearance Is a New Mechanism of Thrombocytopenia. Circ Res. 2023 Oct 27;133(10):826-841. doi: 10.1161/CIRCRESAHA.123.322752. Epub 2023 Oct 26. PMID 37883587